CLINICAL TRIAL: NCT00784199
Title: Validating PROMIS Instruments in Depression
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Duke University (Other); Endeavor Health (Other); University of North Carolina, Chapel Hill (Other); Stanford University (Other); Stony Brook University (Other); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07070241; 5U01AR052155-02 (NIH); 2U01AR052155-06 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2013-05

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Roadmap initiative to develop a computerized system measuring patient-reported outcomes in respondents with a wide range of chronic diseases and demographic characteristics. In the first four years of its existence, the PROMIS network developed item banks for measuring patient-reported outcomes in the areas of pain, fatigue, emotional distress, physical function, and social functioning. During the item banking process, the PROMIS network conducted focus groups, individual cognitive interviews, and lexile (reading level) analyses to refine the meaning, clarity, and literacy demands of all items. The item banks were administered to over 20,000 respondents and calibrated using models based on item response theory (IRT). Using these IRT calibrations, computerized adaptive test (CAT) algorithms were developed and implemented. The network has designed a series of studies using clinical populations to evaluate the item attributes, examine their utility as CATs, and validate the item banks. More information on the PROMIS network can be found at www.nihpromis.org.

DETAILED DESCRIPTION:
In order to validate the item banks and to examine their utility as computerized adaptive tests (CATs), the PROMIS network has designed a series of studies that will allow us to examine the attributes of the measures in "real-world" clinical environments. This protocol is aimed at comparing the psychometric properties of the PROMIS item banks with non-PROMIS "gold standard" instruments currently used in our respective fields (pain and mental health). In this context, note that the proposed study is not intended to evaluate treatment effectiveness, and no control group has been included. The main consideration has been to design a study involving ecologically valid treatments with established efficacy that can be administered and evaluated over the short term (i.e., 3 months). Regardless of their impact in the aggregate, such treatments will generate considerable variability in individual outcomes, and this heterogeneity is optimal for examining relevant psychometric issues. The psychometric issue of greatest concern is the validity of the PROMIS item banks as evidenced in convergent and discriminant validity and responsiveness to change. We also will make initial estimates of clinically significant change as reflected in our PROMIS measures. By combining efforts of the two sites that led in the development of the item banks for emotional distress (University of Pittsburgh) and pain (University of Washington), the study will maximize total sample size and provide a fertile ground for analyses of psychometric functioning of the PROMIS banks.

In addition to psychometric questions, we will also address clinically meaningful questions related to pain, depression, and the relationship between the two. The complex relationship between pain and depression has been observed for years. Both syndromes are mutually exacerbating-pain worsens depression and depression worsens the experience of pain. The domain-related issues of greatest interest focus on the interaction between depression and pain and its impact on treatment outcome (including changes in symptoms of both depression and pain, in acute clinical status, and in social functioning).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Speak, read, and understand English
* Currently in the first 4 months of outpatient treatment at Western Psychiatric Institute and Clinic (WPIC) for major depressive disorder
* Participants will be required to have a minimum score of 12 on the 17-item Hamilton Rating Scale for Depression

Exclusion Criteria:

* Lack of willingness or ability to provide informed consent
* Dementia or other cognitive impairment that would interfere with questionnaire completion
* Lifetime history of any psychotic disorder (e.g., schizophrenia, schizoaffective disorder) or bipolar disorder, as evidenced in the participant's medical records or reported during the Structured Clinical Interview for DSM-IV (SCID)
* Organic affective syndrome (i.e., mood disorder secondary to a general medical condition or substance-induced mood disorder)
* Current psychiatric inpatient treatment
* A history of continuous care for 1 year or more in the mental health care system within the prior 5 years (in order to eliminate patients with more chronic presentations)
* Major medical conditions that influence the central nervous system (e.g., Parkinson's disease, stroke, amyotrophic lateral sclerosis [ALS], multiple sclerosis [MS]), systemic lupus erythematosus [SLE], seizure disorders, etc.)

Note: Persons with common psychiatric comorbidities (e.g., anxiety disorders) will be included. The presence of psychiatric comorbidities will be documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have started treatment for an episode of major depressive disorder in the last 4 months at Western Psychiatric Institute and Clinic (WPIC) in Pittsburgh, PA. WPIC houses the Department of Psychiatry at the University of Pittsburgh Medical Center (UPMC) and serves as the flagship for the UPMC Behavioral Health Network, the psychiatric specialty division of the UPMC Health System. Each year, WPIC provides more than 350,000 patient contacts in its ambulatory care sites.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
PROMIS computerized adaptive tests (CATs) for pain, fatigue, social functioning, depression, anxiety, anger, sleep, wake, and physical functioning, and non-PROMIS measures (conventional instruments) also administered by computer | Assessments at baseline, 1 month, and 3-month follow-up

SECONDARY OUTCOMES:
Judgments of clinically significant change (via diagnostic interviews) and comparison of these changes with the changes reflected in the PROMIS measures | Assessments at baseline, 1 month, and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Pilkonis, PhD, Principal Investigator — University of Pittsburgh